CLINICAL TRIAL: NCT05691920
Title: Ultrasound Guided External Oblique Intercostal Plane Block and Pectointercostal Plane Block for Perioperative Analgesia in Coronary Artery Bypass Graft Surgery: Prospective Randomized Controlled Study
Brief Title: Regional Blocks for CABG Artery Bypass Graft Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305397
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-11

CONDITIONS: Analgesia After Coronary Artery Bypass Graft Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator): Patients will be subjected to bilateral external oblique intercostal plane and pectointercostal plane blocks
  Interventions: Procedure: Pectointercostal plane block and external oblique intercostal plane block
- Opioid group (Active Comparator): Patients will be subjected to fentanyl infusion at a rate of 1μg/kg/h
  Interventions: Procedure: Fentanyl infusion

INTERVENTIONS:
Procedure: Pectointercostal plane block and external oblique intercostal plane block — Patients will be subjected to bilateral external oblique intercostal plane and pectointercostal plane blocks
  Arms: Block group
Procedure: Fentanyl infusion — Patients will be subjected to fentanyl infusion at a rate of 1μg/kg/h
  Arms: Opioid group

SUMMARY:
Pain control after CABG is an essential step to guard against postoperative complications such as lung atelectasis. This major step can be achieved by opioids or regional blocks.

Regional blocks allow better pain control and avoid side effects of opioid based pain control

DETAILED DESCRIPTION:
Ultrasound guided External oblique intercostal plane block and pectointercostal plane block for perioperative analgesia in coronary artery bypass graft surgery: Prospective randomized controlled study

Introduction:

Pain control is a vital component to achieve enhanced recovery after cardiac surgery. Effective postoperative pain control will reduce the incidence of numerous postoperative complications, can facilitate early mobilization and may result in earlier recovery.

Pain control is historically achieved by the administration of opioids, which is associated with well-documented side effects, such as sedation, respiratory depression, pruritus, hallucinations and postoperative nausea and vomiting (PONV). Enhanced recovery following coronary artery bypass grafting (CABG) has gained attention even though there is limited evidence on the efficacy and effectiveness of existing analgesic techniques.

The external oblique intercostal plane and pectointercostal plane blocks are a new modality that will be used to improve pain-related outcomes after CABG surgery, and has not been extensively investigated. Therefore, we will test the hypothesis that external oblique intercostal plane and pectointercostal plane blocks can reduce cumulative opioid consumption for the patients undergoing CABG surgery when added to conventional multi-model intravenous analgesic technique.

The aim of this prospective comparative investigation is to assess the impact of external oblique intercostal plane and pectointercostal plane blocks in a multimodal perioperative analgesic regimen and any related side effects in patients undergoing CABG surgery.

Patients and Methods:

A prospective study will be carried out in Alexandria Main University Hospital on 120 American society of anaesthesiologists (ASA) II, III physical status aged 40-60 years scheduled for major upper abdominal surgery, after approval of the Medical Ethics Committee and an informed written consent. Patients will be categorized into two equal groups, group I (60) will be subjected to bilateral external oblique intercostal plane and pectointercostal plane blocks and group II (60) will be subjected to fentanyl infusion at a rate of 1μg/kg/h. During the patient stay in the ICU, total analgesic requirements will be measured in both groups. Also, sedation level, duration of intubation and length of ICU stay will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CABG surgery

Exclusion Criteria:

* BMI above 40
* allergy for drugs used
* complicated cases
* patient refusal
* chronic opioid use
* cognitive dysfunction
* chronic kidney disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative fentanyl requirements for 24 hours | 24 hours postoperatively
  Visual analogue score will be measured every 2 hours

SECONDARY OUTCOMES:
Visual analogue score | 24 hours postoperatively
  Visual analogue score will be measured every 2 hours
Rescue analgesia | 24 hours postoperatively
  0.5 microgram/kg fentanyl will be given if visual analogue score more than 4
Side effects | 24 hours postoperatively
  Any side effect related to fentanyl or block technique will be detected and treated properly

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request
Supporting Information: Study Protocol, CSR
Time Frame: One year
URL: http://www.alexu.edu.eg

REFERENCES:
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241